CLINICAL TRIAL: NCT03165942
Title: Neuroendocrine Response to Oral Alcohol Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1502015387; 1R21AA025277-01 (NIH); 1K99AA025401-01A1 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Alcoholic Beverages; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alcoholic Beverage (Experimental): Participants will complete an MRI and oral alcohol session.
  Interventions: Other: Alcoholic Beverage; Drug: Ethanol
- Non-Alcoholic Beverage (Placebo Comparator): Participants will complete an MRI and oral non-alcoholic session.
  Interventions: Other: Non-Alcoholic Beverage; Drug: Ethanol

INTERVENTIONS:
Other: Alcoholic Beverage — In addition to the oral delivery, an IV line will be placed for the purpose of drawing blood during the MRI session.
  Arms: Alcoholic Beverage
Other: Non-Alcoholic Beverage — In addition to the oral delivery, an IV line will be placed for the purpose of drawing blood during the MRI session.
  Arms: Non-Alcoholic Beverage
Drug: Ethanol

SUMMARY:
This study proposes to examine both the peripheral and central nervous system responses when light social drinkers and binge/heavy social drinkers are exposed to oral ethanol. The findings will provide a greater understanding of the brain mechanisms (cerebral blood flow and functional connectivity) underlying the association between stress, cortisol release, heart rate variability, alcohol craving, and alcohol stimulant and sedative effects. This knowledge could be significant in developing new therapies for the treatment of alcoholism.

DETAILED DESCRIPTION:
This study was a single-blind, mixed Between Subjects and repeated measures across Alcohol and Placebo conditions in separate sessions in a 2 scan neuroimaging experiment. The two groups of participants were Moderate Social Drinkers and Binge/Heavy Social Drinkers, categorized on the basis of NIAA criteria for moderate non-binge and binge/heavy drinking. Subjects were randomly assigned to receive alcoholic or non-alcoholic beer in scanning condition 1 or condition 2. Before each scan, they were exposed to 3 12 Oz. alcoholic beer or 3 12 Oz. non-alcoholic beer via an Alcohol Taste Test (ATT) during which they were asked to taste the beers to determine if they were same or different. The order of the two conditions was counterbalanced and randomized across participants. Cerebral blood flow (CBF) was then measured using Arterial Spin Labeling. In addition to measuring the different effects of alcoholic beer vs. non-alcoholic beer on CBF, the investigators also measured subjective alcohol effects, alcohol craving, breath alcohol levels, cortisol, and ACTH. Statistical tests were performed to determine if these dependent measures were due to Group, Condition, or a Group x Condition interaction. Finally, the relationship between these variables and the amount of beer consumed at the second post-scan ATT was examined. The post-scan ATT only presented with the choice to drink non-alcoholic beer in order to more clearly predict behavioral motivation for alcohol from PreATT alcohol response in cortisol, CBF and subjective ratings. Data was obtained by research staff, nurse, and MRI technician who were blind to condition as were the subjects but PI and project director were not blind.

ELIGIBILITY:
Inclusion Criteria:

* Binge/Heavy Social Drinkers (HSD): has never met DSM-IV criteria for alcohol or substance dependence; regular alcohol use over the past year of at least 10 drinks per week, including at lease one occasion per week consuming >4 drinks (males) or >3 drinks (females).
* Able to read and write English.
* Light Social Drinkers (LSD): has never met DSM-IV criteria for alcohol or substance dependence; regular alcohol use over the past year of 1-3 drinks per occasion, 1-3 times weekly, with no more than one occasion per month of drinking >4 drinks (male) or >3 drinks (females) (King et al., 2002).
* Do not meet criteria for any Axis I DSM-IV psychiatric diagnoses except for individuals with a past diagnosis of Post-Traumatic Stress Disorder, Major Depressive Disorder, or Obsessive Compulsive Disorder; and provide negative urine toxicology screens during initial appointments and at admission for IV/fMRI sessions.
* Body Mass Index between 20-28.
* No current or former nicotine dependence.

Exclusion Criteria:

* Meet current criteria for dependence on any psychoactive substance, excluding caffeine.
* Current or past history of alcohol dependence or abuse.
* Any current use of opiates or past history of opiate abuse/dependence.
* Current use of any psychoactive drugs, including anxiolytics, antidepressants, naltrexone or antabuse.
* Any psychotic disorder or current psychiatric symptoms requiring specific attention, including need for psychiatric medications for current major depression and anxiety disorders.
* Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, liver, thyroid pathology; subjects on medications for any medical condition will be excluded.
* Peri and post menopausal women, and those with hysterectomies.
* Pregnant and lactating women will be excluded.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Flow | End of Procedure (45 minutes)
  Blood flow is measured in ml/100 grams/minute. The interpretation is that blood flow to that area indicates that region of the brain is responding to the consumption of alcohol or alcohol cues. Change in blood flow will be calculated as the change (and slope) of measurements taken at 10, 20, 30 and 45 minutes during the procedure.
Change in Amount of drink consumed (alcohol or placebo) | Pre-scan ATT and immediately Post scan ATT
  Amount of drink consumed (alcohol or placebo) during the Alcohol Taste Test (ATT)

SECONDARY OUTCOMES:
Changes in Alcohol Effects (BAES) | Post follow up to Procedure (125 minutes)
  Alcohol effects will be measured using the Biphasic Alcohol Effects Scale (BAES). The BAES is a 12 item questionnaire with a 12-120 range. The higher the total value (up to 120), the greater the measured effects of alcohol. The change in alcohol effects will be assessed with the taking the change (and slopes) of measurements at 45, 30 and 5 minutes prior to procedure and comparing it to measurements taken at 65, 95, 110, 125 minutes following the procedure.
Changes in Alcohol Effects (DEQ) | Post follow up to Procedure (125 minutes)
  Alcohol effects will be measured using the Drug Effects Questionnaire (DEQ). The DEQ consists of 5 questions with 5-25 total point distribution. The greater the total points, the greater the measured effect of alcohol. The change in alcohol effects will be assessed with the taking the change (and slopes) of measurements at 45, 30 and 5 minutes prior to procedure and comparing it to measurements taken at 65, 95, 110, 125 minutes following the procedure.
Changes in Alcohol Urges (AUQ) | Post follow up to Procedure (125 minutes)
  The urge to consume alcohol will be measured using the Alcohol Urge Questionnaire (AUQ). The AUQ consists of 8 questions 8-56 total point distribution. The greater the total points, the greater the measured urge to consume alcohol. The change in alcohol urge will be assessed with the taking the change (and slopes) of measurements at 45, 30 and 5 minutes prior to procedure and comparing it to measurements taken at 65, 95, 110, 125 minutes following the procedure.
Change in Cortisol | Post follow up to Procedure (125 minutes)
  The units for cortisol are micrograms/deciliter and the interpretation is that amount has been released into the blood stream from the HPA axis in response to alcohol or alcohol cues. Change in Cortisol will be calculated by taking the change (and slopes) of measurements at 45, 30 and 5 minutes prior to procedure and comparing it to measurements taken at 65, 95, 110, 125 minutes following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Blaine, PhD, Principal Investigator — Addictions, Division of Yale Stress Center; Rajita Sinha, PhD, Principal Investigator — Professor of Psychiatry, Yale Center for Clinical Investigation
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided